CLINICAL TRIAL: NCT04806360
Title: Application of Anterior Spinal Canal Reconstruction and Fusion Surgery for Treating Degenerative Cervical Kyphosis With Stenosis：a Multicenter Randomized Controlled Trial
Brief Title: Anterior Spinal Canal Reconstruction and Fusion Surgery for Treating Degenerative Cervical Kyphosis With Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Naval Specialty Medical Center, China (Unknown); The NO.72 Army Hospital of Huzhou, China (Unknown); 903 Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Xuhua Lu, Director of Traumatic Orthopaedic Department, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020YLCYJ-Y09
Record Dates: First submitted 2021-02-16; First posted 2021-03-19 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Degenerative Cervical Kyphosis With Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACRF group (Experimental): ACRF is a new surgical procedure that previously proposed by our team, it combines the advantages of both the conventional anterior and posterior approach. Eligible patients in this group will receive ACRF surgery.
  Interventions: Procedure: ACRF surgery
- conventional anterior surgery group (Active Comparator): Eligible patients in this group will receive conventional anterior surgery, including anterior cervical discectomy and fusion surgery or anterior cervical corpectomy and fusion surgery.
  Interventions: Procedure: conventional anterior surgery
- conventional posterior surgery group (Active Comparator): Eligible patients in this group will receive conventional posterior surgery, including laminectomy and fusion surgery or laminoplasty surgery.
  Interventions: Procedure: conventional posterior surgery

INTERVENTIONS:
Procedure: ACRF surgery — A new surgical procedure that previously proposed by our team.
  Arms: ACRF group
Procedure: conventional anterior surgery — Anterior cervical discectomy and fusion surgery or anterior cervical corpectomy and fusion surgery.
  Arms: conventional anterior surgery group
Procedure: conventional posterior surgery — Laminectomy and fusion surgery or laminoplasty surgery.
  Arms: conventional posterior surgery group

SUMMARY:
Degenerative cervical kyphosis with stenosis (DCKS) is a common cervical spine degenerative disease, causing pain, numbness, and weakness of limbs, which seriously affect the quality of life of the patient. Surgery is an effective way to treat this condition, however, the best surgical procedure is still controversial. Anterior spinal canal reconstruction and fusion surgery (ACRF) is a new surgical procedure that previously proposed by our team, it combines the advantages of both the conventional anterior and posterior approach. The purpose of this study is to evaluate the safety and effectiveness of ACRF surgery for treating DCKS. A multicenter prospective randomized controlled trial was designed. Eligible patients will be randomly divided into three groups, including the ACRF group, the conventional anterior surgery group, and the conventional posterior surgery group. Demographic data, surgery Information, and follow-up results will be collected and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with degenerative cervical kyphosis with stenosis
* Patients aged between 30 and 70 years
* Patients meet the indications for surgery
* Patients submitted written informed consent

Exclusion Criteria:

* Tumor, infection, or trauma of the cervical spine
* Severe cervical kyphosis that greater than 50°
* Severe ossification of the posterior longitudinal ligament of the cervical spine
* Patients with ankylosing spondylitis
* Previous surgery of the cervical spine

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Japanese Orthopaedic Association Score (JOA) | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Total score 0-17. The lower the score the more severe the deficits.
Change of Neck Disability Index (NDI) | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Ranging from 0%-100%. A higher score indicates more patient-rated disability.
Change of Sagittal Lordosis Angle | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Measured by lateral X-Ray image. The change of lordosis was calculated and compared.
Change of Cross-sectional area of the spinal canal | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Measured by MRI image. The change of cross-sectional area of the spinal canal was calculated and compared.

SECONDARY OUTCOMES:
Reoperation rate | 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Any reoperation involving the same segments or adjacent segments will be calculated.
Change of Pain Scores on the Visual Analog Scale (VAS) | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Ranging from 0-10. A higher score indicates more severe pain.
Change of Range of Motion | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Measured by dynamic X-Ray image.
Complication rate | baseline, 1 month, 3 months, 6 months, 12 months and 24 months post-treatment
  Any complications related to surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Lu, M.D., Principal Investigator — Shanghai Changzheng Hospotal
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided